CLINICAL TRIAL: NCT06893770
Title: Effect of Quran Recital on Quality of Life and Quality of Sleep in Patients Receiving Chemotherapy Due to Breast Cancer
Brief Title: The Effect of the Quran on Quality of Life and Quality of Sleep in Breast Cancer
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ardahan University (Other)
Collaborators: Erzurum Technical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ArdahanU-Simsekli-DS-05
Record Dates: First submitted 2025-03-10; First posted 2025-03-25 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Breast Carcinoma
Keywords: breast cancer; Quran recital; life of quality; sleep of quality
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: randomized controlled design
Who Masked: Participant, Outcomes Assessor
Masking Description: Before the study, a separate consent form was prepared for the experimental group and a separate consent form for the control group, and it was planned to blind the participants by not informing them about which group they were in. In addition, data will be entered with group 1 and group 2 coding for the Quran recital group and the control group, and it was planned to apply statistician blinding.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- experimental group (Experimental): Quran recital
  Interventions: Behavioral: Quran recital
- control group (Active Comparator): standard treatment and care
  Interventions: Other: standard treatment and care

INTERVENTIONS:
Behavioral: Quran recital — standard treatment and care
  Other Names: standard treatment and care
  Arms: experimental group
Other: standard treatment and care — standard treatment and care
  Arms: control group

SUMMARY:
Objective: This study aims to investigate the effects of Quran on quality of life and sleep in patients receiving chemotherapy due to breast cancer.

Method: This study will be conducted with 40 patients with breast cancer receiving chemotherapy at Erzurum City Hospital Outpatient Chemotherapy Unit in a randomized controlled experimental design. Block randomization will be used in group assignment. The breast cancer patient identification form, European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Scale (QLQ-C30) and Pittsburg Sleep Quality Index (PSQI) will be used to collect research data. It is planned to collect research data with a total of four measurements during the application of the first, second, third and last protocols of chemotherapy.

Expected Results: As a result of the study, it is expected that Quran recitation will have a positive effect on quality of life and sleep in patients receiving chemotherapy due to breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Having breast cancer
* Being on chemotherapy
* Being on a chemotherapy protocol every 21 days
* Being over the age of 18
* Not having communication problems
* Being willing to participate in the study

Exclusion Criteria:

* Having a hearing problem
* Having an ear infection or any condition that prevents hearing
* Having other types of cancer other than breast cancer

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-04-15 (Estimated); Primary Completion 2026-04-15 (Estimated); Study Completion 2026-04-15 (Estimated)

PRIMARY OUTCOMES:
The European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Scale (QLQ-C30), Version 3.0 (EORTC QLQ C-30) | From registration to the end of treatment at week 12
  The European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Scale (QLQ-C30), Version 3.0 (EORTC QLQ C-30) will be used to assess quality of life. High general well-being and functional subscale scores indicate high quality of life.

SECONDARY OUTCOMES:
Pittsburg Sleep Quality Index | From registration to the end of treatment at week 12
  The Pittsburgh Sleep Quality Index (PSQI) was used to assess sleep quality. A score of six or above indicates poor sleep quality.

CONTACTS AND LOCATIONS:
Overall Officials: DERYA ŞİMŞEKLİ, Principal Investigator — Ardahan University
Locations (1):
- Erzurum Technical Universitesi, Erzurum, Turkey, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data cannot be shared with third parties in order to protect personal data.